CLINICAL TRIAL: NCT06644885
Title: Complications of the Cephalic Route in Implantable Site Placement in Children
Acronym: SitePedia
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC24_0097
Record Dates: First submitted 2024-10-04; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Surgical Complications; Device Safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with TIVAD
  Interventions: Procedure: TIVAD implantation complications

INTERVENTIONS:
Procedure: TIVAD implantation complications — Follow up and post operative outcome of patients with devices implantation

SUMMARY:
Totally implantable venous access devices (TIVADs) offer long-term central venous access for children requiring intravenous treatments. Their use is recommended in infants (31 days - 1 year old) for >31 days of non-peripherally compatible therapy, and in children and adolescents (>1 year old) for any intravenous therapy lasting more than 31 days. Indications include chemotherapy administration and chronic disease management, avoiding repeated peripheral venous punctures and causing less interference with the activities of the patients.

There are several methods for TIVAD placement, but the optimal evidence-based method remains unclear . The two main approaches for TIVAD placement are closed cannulation of a vein, followed by insertion of the catheter in Seldinger technique, and the surgical insertion of the catheter into a vein through an open cut-down technique 5-7. Different location of insertion are possible: by closed cannulation, the catheter is usually placed in subclavian vein, internal jugular vein, and brachiocephalic vein; by open cut-down it can be placed in external jugular vein, axillary vein, or cephalic vein.

Thanks to progress in medical and surgical care, children are nowadays surviving previously fatal illnesses, but with the need of long-term treatments. For this reason, it's essential to preserve their vessel health. With this objective, in the CHU of Angers, physicians prefer trying first the cephalic vein cutdown for TIVAD positioning in children, reserving the use of other venous accesses in case of failure of this procedure or the need for multiple devices implantations.

To date, few reports have been published about cephalic vein cutdown in children. It is a common opinion that this technique can't be successfully performed in patients under a certain limit of weight or age. In this context, the investigators conducted a retrospective single-centre study to analyse the results of cephalic vein cutdown in children. The primary aim was to describe the feasibility of this technique in paediatric population and identify the risks factors associated with its failure. In addition, this study describes indications, outcomes, and complications of TIVAD implantation.

ELIGIBILITY:
Inclusion Criteria:

* All patients under 18 years who underwent TIVAD implantation between 2012 and 2022.
* Patients for whom cephalic vein cutdown was the first attempted surgical technique for device placement.

Exclusion Criteria:

* Patients who previously had a central venous access

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients operated in the CHU of Angers
Sampling Method: Non-Probability Sample
Enrollment: 426 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Characteristics of the study group | 1 year
  Risk factors for cephalic vein cutdown failure for TIVAD positioning

SECONDARY OUTCOMES:
cephalic vein cutdown | 1 year
  Post-operative complications of cephalic vein cutdown
Post-operative complications | 1 year
TIVAD removal | 1 year